CLINICAL TRIAL: NCT02383342
Title: Development of Postoperative Pain; Clinical and Genetic Factors
Brief Title: Pain Predict Genetics
Acronym: PPG
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL26908.091.12
Record Dates: First submitted 2015-01-28; First posted 2015-03-09 (Estimated); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Chronic Pain; Acute Pain
Keywords: Clinical predictors; Genetic Factors
MeSH Terms: conditions — Chronic Pain; Acute Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood for DNA
Oversight: Data Monitoring Committee: Yes | US Export: No

SUMMARY:
Pain is the most frequent cause of suffering and disability in society. Despite considerable involvement of genetic factors in pain sensation and sensitivity, the individual genes involved remain largely unidentified.

In this project the investigators will follow patients undergoing elective major surgery for the development of acute and chronic pain. The investigators will search for clinical as well as genetic factors that can predict the development of pain. These can serve as biomarkers to predict acute and chronic pain development and progression in individual patients and help early individual treatment adaptation.

DETAILED DESCRIPTION:
Pain is the most frequent cause of suffering and disability in society. Chronic pain seriously impairs quality of life of millions of people worldwide. 10-50% of surgical patients report chronic pain after surgery; up to 10% report severe pain. Thus, chronic pain is a significant medical and financial burden to society.

Despite considerable involvement of genetic factors in pain sensation and sensitivity, individual genes involved remain largely unidentified. Knowledge of genetic factors, their phenotypic expression in pain processing, and their link to neuronal correlates can improve understanding of pain aetiology and processes involved in pain perception and chronification. Also, they can serve as biomarkers to predict chronic pain development and progression in patients and help early individual treatment adaptation.

In this study the investigators will establish a prospective database and biobank of patients undergoing elective major surgery. Using data from the database and biobank, the investigators will identify genetic factors contributing to development of acute and chronic pain after surgery.

Over a period of 10 years the investigators will prospectively include up to 10,000 patients visiting the hospital for elective major surgery. Data defining participants demographics, medical history and questionnaire data will be collected and stored in dedicated databases. Additional details (surgery and perioperative management, pain processing phenotypes and surgical and pain outcomes) will be stored.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Ages 18 - 80 years, consenting, planned surgery, able to understand and answer questionnaires.

Exclusion Criteria:

* Non-consent, inability to give consent, unplanned and emergency surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing elective major surgery at Radboud university medical center (Nijmegen, The Netherlands) Patients will be recruited prospectively and consecutively via the anaesthetic preoperative outpatients' clinic.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-05-12 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Genetic risk factors for the development of acute pain using a visual analogue scale. | 7 days
  All patients will be followed for 1 year after elective surgery, during this period the investigators will collect acute pain measures using a visual analogue scale (ranging from 0 (no pain) -10 (pain)) before the operation and 1, 2, 3 and 7 days after the operation.
Genetic risk factors for the development of chronic pain (defined as pain (yes or no) for more than 3 months in one specific body area). | 6 months
  All patients will be followed for 1 year after elective surgery, during this period the investigators will collect chronic pain measures using a questionnaire before the operation and 1 week, 3 months and 6 months. Chronic pain is defined as pain at a specific body side (yes/no) for more than 3 months.

SECONDARY OUTCOMES:
If the pain influences daily functioning will be assesed with the pain disability index. | 6 months
  The pain disability index will be used to assess whether the observed acute or chronic pain influences daily life. The pain disability index will be collected before the operation and at week 1, 3 months and 6 months.
Is fear before an operation related to the development of acute and chronic pain after the operation. | once pre-operatively
  The Amsterdam Preoperative Fear and Information Scale (APAIS)(Moerman et al. Anesth Analg. 1996 Mar;82(3):445-51) will be used to assess whether the observed acute or chronic pain can be linked to fear before an operation. The measure will be collected before the operation. The scores on the anxiety scale of the APAIS range from 4 (not anxious) to 20 (highly anxious). And the scores on the information scale of the APAIS range from 2 (no need for information) to 10 (high need for information).
Is the Pain Catastrophizing Scale related to the development of acute and chronic pain after the operation. | once pre-operatively
  The Pain Catastrophizing Scale (Sullivan et al. Psychol Assess 1995;7:524-32) will be used to assess whether the observed acute or chronic pain are association with the Pain Catastrophizing Scale. The Pain Catastrophizing Scale contains 13 items (all items are rated on a 5 point scale). The measure will be collected before the operation.
Is Pain Sensitivity related to the development of acute and chronic pain after the operation. | once pre-operatively
  The Pain Sensitivity Questionnaire (PSQ; Ruscheweyh et al.Pain. 2009 Nov;146(1-2):65-74) will be used to assess whether the observed acute or chronic pain are association with a higher pain sensitivity. This questionnaire consists of 17 questions, each describing a daily life situation on a numeric rating scale ranging from 0 (not painful at all) to 10 (worst pain imaginable). The pain sensitivity questionnaire will be collected before the operation.
Is the size of the incision made during the operation associated with pain development. | 6 months
  The incision size will be measured and reported by the patients to investigate whether this is linked to the development of acute or chronic pain
Is days in hospital after the operation associated with pain development. | 6 months
  Number of days in the hospital will be recorded to investigate whether this is linked to the development of acute or chronic pain.
Is medication use after the operation assocaited with pain development. | 6 months
  Type of (pain)medication and duration of medication use will be recorded by questionnaires and electronic health records. The investigators will analyse if medication type or duration of medication use is associated with pain development.

CONTACTS AND LOCATIONS:
Overall Officials: Han G Brunner, Prof. PhD., Study Director — Radboud University Medical Center; Barbara Franke, Prof. PhD., Principal Investigator — Radboud University Medical Center; Gert Jan Scheffer, Prof. PhD., Study Chair — Radboud University Medical Center; Rianne van Boekel, PhD., Principal Investigator — Radboud University Medical Center; Kris Vissers, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands

REFERENCES:
- [Derived] Li S, van Boekel RLM, van den Heuvel SAS, Coenen MJH, Vissers KCP. Pain predict genetics: protocol for a prospective observational study of clinical and genetic factors to predict the development of postoperative pain. BMJ Open. 2022 Nov 29;12(11):e066134. doi: 10.1136/bmjopen-2022-066134. PMID 36446453